CLINICAL TRIAL: NCT02583360
Title: Neonatal Esophagus and Airway Interactions in Health and Disease
Brief Title: Mechanisms and Management of Infant Dysphagia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sudarshan Jadcherla (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Ohio State University (Other); Medical College of Wisconsin (Other)
Responsible Party: Sponsor-Investigator, Sudarshan Jadcherla, Principal Investigator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-00794; P01DK068051 (NIH)
Record Dates: First submitted 2015-10-20; First posted 2015-10-22 (Estimated); Results first posted 2020-12-16 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Dysphagia; Airway Aspiration; Airway Penetration
Keywords: Infant; Feeding difficulties; Dysphagia
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: Eligible consented subjects (study) from a single center will undergo standard of care diagnostic VFSS in combination with the research intervention of utilizing manometry procedures to measure pharyngo-esophageal motility to aid with precise diagnosis, either concurrent or sequential. They will then have parental choice of preferred feeding therapy based on combined testing methods rather than therapy being prescribed by the VFSS results. The controls are those who had VFSS alone (standard of care) with treatment based solely on VFSS guided provider recommendations from the same single center.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study (Active Comparator): Eligible subjects (study) will undergo diagnostic VFSS in combination with manometry, either concurrent or sequential. They will have parental choice of preferred feeding therapy.
  Interventions: Diagnostic Test: Combined testing (diagnostic VFSS + research HRM) + Parent Preferred Therapy
- Control (No Intervention): Eligible subjects who had VFSS alone with provider recommendations from the same single center.

INTERVENTIONS:
Diagnostic Test: Combined testing (diagnostic VFSS + research HRM) + Parent Preferred Therapy — Addition of research HRM along with diagnostic VFSS with parental choice of therapy
  Arms: Study

SUMMARY:
The purpose of the investigator's study is to evaluate the causes of feeding difficulty in infants. New treatments can be possible only if the cause is known. In this study, the investigator plans to evaluate the movement of the muscles in an infant's mouth, throat (pharynx) and food pipe (esophagus) that are responsible for moving the food down into the stomach and that help protect an infants airway.

DETAILED DESCRIPTION:
Infants with chronic feeding difficulties exhibit inadequacy of suck-swallow and breathe coordination, regurgitation or vomiting, gastroesophageal reflux disease, and airway aspiration. Often these infants must rely on feeding tubes, either inserted through the nose or surgically placed, to meet their nutrition and hydration needs until they are able to orally feed safely, effectively, and efficiently. The process of assessment and treatment of swallowing disorders is often stressful for the infants and their providers, including parents. The goal of this study is to combine two commonly used diagnostic techniques (video fluoroscopy swallow studies and esophageal manometry) to more comprehensively evaluate feeding from the mouth to the stomach in infants. The hope is that by doing so treatment strategies can be improved.

: Eligible subjects (study) will undergo diagnostic VFSS in combination with manometry, either concurrent or sequential. They will have parental choice of preferred feeding therapy. The data is from single center prospective observational study. The controls are those who had VFSS alone with provider recommendations from the same single center.

In addition, we are also embarking on alternate strategies to achieve the original stated aims: 1) Mechanisms of dysphagia is ascertained by studying concurrent recordings of VFSS and manometry. 2) Feeding outcomes of Dysphagic infants are ascertained by evaluating the discharge outcomes and 1-year feeding outcomes among those that had evaluation of dysphagia using VFSS. 3) Dysphagic infants that had sequential VFSS and manometry studies are evaluated to test which method is a better predictor of stated outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Infants with feeding-related aero-digestive symptoms
* ≤60 weeks PMA (both pre-term and full term)
* History of orally feeding ≥ 25% of least 50% of prescribed feeding volume
* Room air or supplemental oxygen of ≤1liter/minute (LPM)

Exclusion Criteria:

* Direct breast feeding exclusively
* Known genetic, metabolic or syndromic disease
* Neurological diseases such as Grade 3 or 4 intraventricular hemorrhage (IVH) or intracranial hemorrhage (ICH), moderate to severe perinatal asphyxia or stroke
* Craniofacial, airway or foregut malformations
* History of craniofacial, foregut, ears, nose and throat (ENT) or neurosurgery

Ages: 38 Weeks to 60 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 109 (Actual)
Dates: Start 2015-10-02 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sudarshan R Jadcherla, MD, Principal Investigator — The Research Institute at Nationwide Children's Hospital; Reza Shaker, MD, Study Chair — Medical College of Wisconsin
Locations (1):
- The Research Institute at Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jadcherla SR, Stoner E, Gupta A, Bates DG, Fernandez S, Di Lorenzo C, Linscheid T. Evaluation and management of neonatal dysphagia: impact of pharyngoesophageal motility studies and multidisciplinary feeding strategy. J Pediatr Gastroenterol Nutr. 2009 Feb;48(2):186-92. doi: 10.1097/MPG.0b013e3181752ce7. PMID 19179881
- [Background] Jadcherla SR, Peng J, Moore R, Saavedra J, Shepherd E, Fernandez S, Erdman SH, DiLorenzo C. Impact of personalized feeding program in 100 NICU infants: pathophysiology-based approach for better outcomes. J Pediatr Gastroenterol Nutr. 2012 Jan;54(1):62-70. doi: 10.1097/MPG.0b013e3182288766. PMID 21694638
- [Background] Jadcherla SR, Gupta A, Stoner E, Fernandez S, Shaker R. Pharyngeal swallowing: defining pharyngeal and upper esophageal sphincter relationships in human neonates. J Pediatr. 2007 Dec;151(6):597-603. doi: 10.1016/j.jpeds.2007.04.042. Epub 2007 Aug 23. PMID 18035137
- [Background] Jadcherla SR, Shubert TR, Gulati IK, Jensen PS, Wei L, Shaker R. Upper and lower esophageal sphincter kinetics are modified during maturation: effect of pharyngeal stimulus in premature infants. Pediatr Res. 2015 Jan;77(1-1):99-106. doi: 10.1038/pr.2014.147. Epub 2014 Oct 3. PMID 25279989

RESULTS

PARTICIPANT FLOW:
Groups:
- Study: Eligible subjects (study) will undergo diagnostic VFSS in combination with manometry, either concurrent or sequential. They will have parental choice of preferred feeding therapy.
  Combined Diagnostic testing (VFSS + HRM) + Parent Preferred Therapy: HRM along with diagnostic VFSS with parental choice of therapy
Period: Overall Study
Arm/Group | Study | Control
Started | 60 | 49
Completed | 60 | 49
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Study | Control | Total
Number analyzed (Participants) | 60 | 49 | 109
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 60 | 49 | 109
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: weeks] — Postmenstrual age at time of study
  weeks | 45.7 [36.4 to 60.7] | 45.7 [38.4 to 57] | 45.7 [36.4 to 60.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 30 | 56
  Male | 34 | 19 | 53
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 15 | 24
  White | 50 | 31 | 81
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 60 | 49 | 109

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Safe Oral Feeding
Description: The primary endpoint is the feeding success defined as full oral feeding (no tube feeds feeds) without symptoms that require interventions
Time Frame: Up to 4 weeks after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Study | Control
Number analyzed (Participants) | 60 | 49
Participants | 51 | 31
Statistical Analysis 1: Comparison: Study vs Control; Test type: Superiority; p = 0.008, Chi-squared

2. Secondary Outcome: Weight Growth Velocity in Grams/Day
Description: The investigators will measure and track growth velocity (grams/day) during this time period. This will be completed through chart reviews of weight from subsequent clinic visits and parent interviews.
Time Frame: 4 weeks
Population: Unable to get growth velocity on all patients as they were not all hospitalized or weight at 4 weeks after study
Measure: Mean (Standard Deviation); unit: grams/day
Arm/Group | Study | Control
Number analyzed (Participants) | 27 | 46
grams/day | 27 (11.1) | 26.7 (11.5)
Statistical Analysis 1: Comparison: Study vs Control; Test type: Superiority; p = 0.907, t-test, 2 sided

3. Secondary Outcome: Hospital Length of Stay From Admission to Discharge in Days
Description: The investigators will track the subjects length of hospitalization which included their initial study procedure.
Time Frame: from hospital admission until discharge
Population: Some patients in study group were outpatient
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Study | Control
Number analyzed (Participants) | 38 | 49
days | 43.6 (49.7) | 49.9 (58.4)
Statistical Analysis 1: Comparison: Study vs Control; Test type: Superiority; p = 0.592, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Study | Control
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/49
Other Adverse Events (participants affected / at risk) | 0/60 | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-02): https://cdn.clinicaltrials.gov/large-docs/60/NCT02583360/Prot_SAP_000.pdf